CLINICAL TRIAL: NCT05508321
Title: Nasal Brushing for the Diagnosis and Understanding of Telomeropathies
Acronym: TELOSTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/07FEV/046
Record Dates: First submitted 2022-08-10; First posted 2022-08-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Telomere Disease; Telomere Shortening
Keywords: telomere; cellular senescence; smell
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Intervention Model Description: Prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with confirmed or suspected telomeropathy (Experimental): Patients with idiopathic pulmonary fibrosis, adult or pediatric medullar dysplasia or myelodysplasia, unexplained liver cirrhosis or unexplained liver regenerative nodular hyperplasia.
  Interventions: Diagnostic Test: Nasal brushing; Diagnostic Test: Sniffin' Sticks
- Controls (Other): Age and sex-matched control participants
  Interventions: Diagnostic Test: Nasal brushing; Diagnostic Test: Sniffin' Sticks

INTERVENTIONS:
Diagnostic Test: Nasal brushing — Nasal brushing to harvest nasal cells and perform staining experiments
Diagnostic Test: Sniffin' Sticks — Assessment of olfactory function

SUMMARY:
To date, the diagnosis of telomeropathies is based on telomere length measured in blood cells. However, this type of analysis is not always sufficient because some mutations underlying the development of telomeropathies are not associated with abnormal shortened telomeres. Since telomere dysfunction analysis cannot be performed on blood cells, it is mandatory to have access to another cellular material. To date, skin biopsies are performed to obtain fibroblasts. However, this technique is relatively invasive. The aim of this project is to assess whether nasal epithelial cells obtained through nasal brushing could offer the opportunity to detect cellular alterations and mutations involved in telomeropathies, in a mildly invasive way. If successful, this technique could become a non-invasive clinical tool for the diagnosis work-up of telomeropathies. Moreover, investigators aim to assess whether olfactory function is impaired in patients with telomeropathies.

DETAILED DESCRIPTION:
Endpoint #1: To assess the suitability of nasal brushing analyses for the diagnosis of telomeropathies.

To date, the complete diagnosis of telomeropathies, including the identification of responsible mutations, is based on blood samples and fibroblast cultures obtained through skin biopsies. Cells obtained through nasal brushing offer the opportunity to detect cellular alterations and mutations involved in telomeropathies, in a mildly invasive way. Investigators will thus assess a population of patients with a suspicion of telomeropathy, using a nasal brushing, and will compare their nasal brushing results to those of age-matched healthy controls. In patients, results of nasal brushing will be compared to standard of care blood test (leukocyte telomere length using Flow-FISH technique). If investigators confirm that the nasal brushing offers the opportunity to i) detect damaged telomeres and premature cellular senescence and ii) identify mutations related to telomeropathies, this technique could become a non-invasive clinical tool for the diagnosis work-up of telomeropathies.

Endpoint #2: To develop primary cell cultures for the functional study of new germline mutations.

To date, various germline mutations have already been identified in telomeropathy patients, in a total of 17 genes. Understanding how these mutations were affecting telomere biology relied on in vitro studies with either patient-derived fibroblasts or engineered human cell lines recapitulating the mutation. This was a mandatory step towards the molecular understanding of these pathologies. Because olfactory neural precursors have the capacity to grow in culture, this offers the additional possibility to perform functional studies on primary cultures of nasal brushing-derived cells for novel mutations, with still unknown impact on telomeres, that would be identified. Again, this could advantageously replace patients' fibroblast cultures established through skin biopsy.

Endpoint #3: To evaluate whether patients with telomeropathies have impaired olfactory function.

Olfactory function is decreased in several diseases and is increasingly recognized as an indicator of biological aging. To date, no data exist regarding the impact of telomeropathies on olfactory function. Therefore, investigators aim to psychophysically assess olfactory function in patients with telomeropathies, in comparison to age-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients : Having a suspicion of or a confirmed telomeropathy

Exclusion Criteria:

Patients and controls:No access to the olfactory cleft Patients and controls: Abnormal endoscopic finding (i.e. meningocele, vascular ectasia)

Specific exclusion criteria for smell assessment (outcome 3):

Patients and controls: History of neurological or psychiatric disorder known to interfere with olfactory function or olfactory trouble (postinfectious, posttraumatic, toxic) Patients and controls: History of chronic rhinosinusitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the suitability of nasal brushing analysis for the diagnosis of telomeropathies through evaluation of cellular senescence (SA-B-gal activity) and damaged telomeres (FISH/IF) | 5 minutes
  Investigators will evaluate if it is possible to detect damaged telomeres (via FISH/IF - Fluorescence In Situ Hybridation /ImmunoFluoresence -) and premature cellular senescence in patients (via SA-B-gal activity - Senescence Associated Beta-galactosidase activity measurement - and senescence associated biomarkers by qRT-PCR - quantitative Reverse Transcription - Polymerase Chain Reaction - ), in comparison to healthy controls.

SECONDARY OUTCOMES:
To develop primary cell cultures to study how the germline mutation affects telomere integrity in vitro through functional telomere assays | 5 minutes
  Cells harvested from the nasal mucosa will be cultived and analysed to detect telomeric DNA damage and premature cellular senescence

OTHER OUTCOMES:
To assess whether patients with telomeropathies have impaired olfactory function | 20 minutes
  Olfactory function will be assessed using the validated Sniffin' Sticks test

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Huart, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clinique Universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT05508321/Prot_SAP_000.pdf